CLINICAL TRIAL: NCT06558838
Title: A Randomized, Parallel Group, Pilot Study to Assess Efficacy and Safety of Acyclovir-penciclovir Cream Versus an Active Comparator (Abreva) in the Suppression of Herpes Simplex Virus Eruptions in Subjects With a History of Herpes Labialis
Brief Title: Efficacy and Safety of Acyclovir-penciclovir Cream Versus an Abreva in the Suppression of Herpes Simplex Virus Eruptions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Hull, Professor, Dermatology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00143253
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Herpes Simplex Oral
MeSH Terms: conditions — Stomatitis, Herpetic | interventions — docosanol

STUDY DESIGN:
Intervention Model Description: This will be a randomized, efficacy assessor-blinded, parallel group, pilot study.
Who Masked: Outcomes Assessor
Masking Description: Efficacy assessments will be done by a qualified trained blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (acyclovir-penciclovir cream) (Experimental): Patients will treat herpes simplex eruption with active study drug.
  Interventions: Drug: acyclovir-penciclovir cream
- Active Comparator (Abreva) (Active Comparator): Patients will treat herpes simplex eruption with Abreva.
  Interventions: Drug: Abreva

INTERVENTIONS:
Drug: acyclovir-penciclovir cream — Patients will treat their cold sore with active study drug based upon their randomization
  Arms: Study Drug (acyclovir-penciclovir cream)
Drug: Abreva — Patients will treat their cold sore with Abreva based upon their randomization
  Other Names: Docosanol
  Arms: Active Comparator (Abreva)

SUMMARY:
This will be a randomized, efficacy assessor-blinded, parallel group, pilot study of up to 40 subjects with documented herpes labialis. Patients will be treated with the study drug, acyclovir-penciclovir cream, or the active comparator of Abreva.

Potential subjects will be assessed during a screening visit that must take place no greater than 2 weeks prior to the Day 1 (Baseline) visit. During the screening period, subjects that meet all other entry criteria will undergo Ultraviolet susceptibility testing to determine the subject's individual minimal erythema dose (MED). Ultraviolet susceptibility testing takes place over two days with exposure to Ultraviolet light on specified regions on the subject's back followed by an assessment of the exposed areas 24 hours later to identify the MED. Subjects who have a measurable MED will be allowed to enroll in the study. Each subject will be randomly assigned in a 1:1 ratio to receive either acyclovir-penciclovir cream or Comparator (Abreva).

Patients who express a cold sore will track the lesion with a diary card to rate their pain levels, and any unusual symptoms at Day 1, Day 3, Day 5, Day 7, and Day 10. Patients may also take photographs of the lesion throughout the study.

DETAILED DESCRIPTION:
This will be a randomized, efficacy assessor-blinded, parallel group, pilot study of up to 40 subjects with documented herpes labialis.

Potential subjects will be assessed during a screening visit that must take place no greater than 2 weeks prior to the lesion induction visit. During the screening period, subjects that meet all other entry criteria will undergo ultraviolet (UV) susceptibility testing to determine their individual minimal erythemal dose (MED). UV susceptibility testing takes place over two days with exposure to UV light on specified regions on the subject's back followed by an assessment of the exposed areas 24 hours later to identify the MED. Subjects who have a measurable MED will be allowed to continue to the induction visit. Patients that do not have measurable MED response will be considered screen failures or patients may have repeat MED testing with different levels.

At the Induction Visit, subjects will undergo UV radiation at a level 3 times their MED. The exposed area of the lip will be marked with indelible ink and a baseline photo may be taken. Each subject will then be randomly assigned in a 1:1 ratio to receive either acyclovir-penciclovir cream or Comparator. Subjects will be dispensed study medication and instructed how to apply it to the exposed area. When the patient first senses the start of developing a cold sore and applies study medication will be considered Day 1. Dosing of the study product will be done five times daily, beginning at the time that a subject first senses the start of the prodromal phase (Day 1). Subjects will be given a diary card to record their pain levels, progression of lesion development and any unusual symptoms (not normally seen with their outbreaks).

Patients will be called daily by the study team after their induction visit to determine the start of prodrome. If after 7 days, the patient does not develop any prodromal senses, the patient will be considered an induction failure.

When the patient first senses signs or symptoms of a cold sore, the patient will have the Day 1 visit conducted within 24 hours. Day 1 visit may be conducted in person or as a MyChart Virtual Visit. Patient's diary card will be reviewed and if the patient have experienced a prodrome and/or lesion since the induction visit, their compliance with dosing will be checked. If the subject has noted any unusual symptoms, these will be discussed with medical personnel to determine if the symptoms represent a treatment emergent adverse event (AE). A photo will be taken of the irradiated area (as marked at the induction visit). The blinded assessor will assess the prodrome and/or lesion and take measurements.

On Days 3, 5, and 7, the subject will return to the clinic or follow up via virtual video call for assessment of the irradiated area. Study staff will review the subject diary to determine if the subject is correctly noting the lesion stage. Subjects will have a photo taken of the radiated area and asked to continue with dosing as instructed. Any diary card notation of unusual symptoms in subjects will be reviewed by study staff to determine if the symptoms represent a treatment emergent adverse event. The blinded assessor will assess the prodrome and/or lesion and take measurements. More study product may be dispensed as needed. Most subjects' lesions will have resolved by day 7, and those subjects will end study treatment after 7 full days of treatment. If lesion has not resolved by day 7, the maximum number of days the patient may use study drug treatment is 10 days.

The End of Study (EOS) is the final study visit that will take place on Day 10. A photo will be taken of the irradiated area, the diary card will be carefully reviewed and study product (including empty containers) will be collected. If subjects reach EOS without full resolution of their lesion(s), those subjects will discuss treatment options with the study doctor for remainder of the outbreak.

Measurements will be taken. If an adverse event has occurred but has not resolved by the EOS visit, the subject will be contacted once weekly and status noted until such time as the event has resolved. The blinded assessor will assess the prodrome and/or lesion.

A Safety follow-up phone call will occur 2 days after the EOS to determine if any new adverse events have occurred.

ELIGIBILITY:
Inclusion Criteria:

* Understands the requirements of the study and provides written informed consent prior to undergoing any study-related procedures.
* Subject is a male or female between the ages of 18-80 years old, inclusive.
* Fitzpatrick skin type II or III.
* History of at least one year of herpes labialis induced by UV exposure.
* Able to recall exact location of most common or most recent outbreak.
* History of at least 50% of cold sore outbreaks occurring with UV (sun) exposure.
* At least 1 HSV-1 outbreak within the past 12 months.
* Experiences prodromal symptoms before HSV-1 outbreaks.
* Subject is willing and able to comply with protocol-specified dosing, visits to the clinic and tracking of pain.

Exclusion Criteria:

* Outbreak <2 weeks prior to enrollment.
* History of herpes simplex vaccine.
* On antiviral suppression within the past 30 days.
* Requires more than acetaminophen for pain from recurrent HSV outbreaks.
* On any systemic or topical steroid, immune suppressant or chemotherapeutic agent within the past 14 days.
* Use of tanning beds, history of sunburn, or beach vacation <2 weeks prior to enrollment.
* History of photosensitivity, lupus erythematosus, or current use of a highly photosensitizing medication in the opinion of the investigator.
* Current immunosuppressed state due to underlying disease (i.e. HIV infection) concomitant treatment (i.e. chemotherapy).
* Current upper respiratory tract infection or any active illness that could trigger cold sores or affect overall health of the patient or the assessment of the study agent.
* Pregnant or intending to become pregnant during the study.
* Abnormal skin conditions in the area of the recurrent HSV1 outbreaks.
* Enrolled in another clinical trial within the past 30 days.
* On any analgesics or NSAIDs that cannot be stopped during the study.
* Alcohol or drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects using acyclovir-penciclovir cream versus those using the Comparator, who do not progress to Stage 3 (vesicle) of a herpes labialis outbreak following UV radiation exposure | up to 25 days per patient
  We will measure the number of subjects who do not progress to Stage 3 of herpes labialis outbreak

SECONDARY OUTCOMES:
Time of duration of the lesion until healed (loss of hard crust) of patients using acyclovir-penciclovir cream compared to those using the active comparator. | up to 25 days per patient
  We will measure the number of days lesions take to heal of patients using EDTA eye drops compared to those using the active comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Hull, M.D., Principal Investigator — University of Utah Dermatology
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheshenko N, Trepanier JB, Gonzalez PA, Eugenin EA, Jacobs WR Jr, Herold BC. Herpes simplex virus type 2 glycoprotein H interacts with integrin alphavbeta3 to facilitate viral entry and calcium signaling in human genital tract epithelial cells. J Virol. 2014 Sep 1;88(17):10026-38. doi: 10.1128/JVI.00725-14. Epub 2014 Jun 18. PMID 24942591
- [Background] Evans TG, Bernstein DI, Raborn GW, Harmenberg J, Kowalski J, Spruance SL. Double-blind, randomized, placebo-controlled study of topical 5% acyclovir-1% hydrocortisone cream (ME-609) for treatment of UV radiation-induced herpes labialis. Antimicrob Agents Chemother. 2002 Jun;46(6):1870-4. doi: 10.1128/AAC.46.6.1870-1874.2002. PMID 12019102
- [Background] Hunsperger EA, Wilcox CL. Capsaicin-induced reactivation of latent herpes simplex virus type 1 in sensory neurons in culture. J Gen Virol. 2003 May;84(Pt 5):1071-1078. doi: 10.1099/vir.0.18828-0. PMID 12692270
- [Background] Jensen LA, Hoehns JD, Squires CL. Oral antivirals for the acute treatment of recurrent herpes labialis. Ann Pharmacother. 2004 Apr;38(4):705-9. doi: 10.1345/aph.1D285. Epub 2004 Feb 13. PMID 14966254
- [Background] Raborn GW, Grace MG. Recurrent herpes simplex labialis: selected therapeutic options. J Can Dent Assoc. 2003 Sep;69(8):498-503. PMID 12954137
- [Background] Spruance SL. The natural history of recurrent oral-facial herpes simplex virus infection. Semin Dermatol. 1992 Sep;11(3):200-6. PMID 1390034
- [Background] Spruance SL, Rowe NH, Raborn GW, Thibodeau EA, D'Ambrosio JA, Bernstein DI. Peroral famciclovir in the treatment of experimental ultraviolet radiation-induced herpes simplex labialis: A double-blind, dose-ranging, placebo-controlled, multicenter trial. J Infect Dis. 1999 Feb;179(2):303-10. doi: 10.1086/314605. PMID 9878012
- [Background] Spruance SL, McKeough MB. Combination treatment with famciclovir and a topical corticosteroid gel versus famciclovir alone for experimental ultraviolet radiation-induced herpes simplex labialis: a pilot study. J Infect Dis. 2000 Jun;181(6):1906-10. doi: 10.1086/315528. Epub 2000 May 31. PMID 10837169